CLINICAL TRIAL: NCT04953156
Title: A Comparative Study Between Nitroglycerine Infusion and Dexmedetomidine Infusion in Intraoperative Management of Uncontrolled Hypertension
Brief Title: Nitroglycerine Versus Dexmedetomidine Infusion in Intraoperative Management of Uncontrolled Hypertension
Status: Completed | Type: Observational
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Lecturer of Anesthesia and Pain management, National Cancer Institute, Egypt
Other Study IDs: AP2105-50107
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nitroglycerin; Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nitroglycerin: data of patients meeting the eligibility criteria and received nitroglycerine infusion will be retrieved from medical records.
  Interventions: Drug: Nitroglycerin
- Dexmedetomidine: patients will receive dexmedetomidine bolus dose of 1 mic/kg over 20 minutes followed by intravenous infusion of 0.2-0.7 mic/kg/hr adjusted according to each patient hemodynamic response
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Nitroglycerin — data will be retrieved from intraoperative medical records for the period from May 2020 to May 2021 for patients meeting the eligibility criteria who developed uncontrolled elevation of their blood pressure and received nitroglycerine infusion
  Groups: Nitroglycerin
Drug: Dexmedetomidine — All patients who develop uncontrolled elevation of their blood pressure and meeting the eligibility criteria from July 2021 to July 2022 will receive dexmedetomidine bolus of 1mic/kg over 20 minutes and then continuous infusion of 0.2-0.7 mic/kg/hour adjusted according to each patient hemodynamic response.
  Groups: Dexmedetomidine

SUMMARY:
This study aim to compare the efficacy of intraoperative dexmedetomidine infusion versus Nitroglycerin infusion in cancer patients with accidental uncontrolled intraoperative elevation of blood pressure.

DETAILED DESCRIPTION:
Nitroglycerine is a direct vessel wall vasodilator with more venodilator effect than arterial dilator effect. It is used as an anti-anginal and antihypertensive drug. On the other hand, dexmedetomidine is a highly selective alpha 2 adrenergic agonist with sympatholytic effect. This study aim to compare the efficacy of intraoperative dexmedetomidine infusion versus Nitroglycerin infusion in cancer patients with accidental uncontrolled intraoperative elevation of blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients with controlled hypertension and undergoing surgical procedures under general anesthesia
* ≥ Age 18 years.

Exclusion Criteria:

* patient refusal
* patients on Beta blockers
* kidney or liver function impairment
* bradycardia, any degree of heart block and severe cardiorespiratory disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with controlled hypertension and undergoing surgical procedures under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood pressure values | Intraoperative period
  measurements of blood pressure

SECONDARY OUTCOMES:
Intraoperative heart rate values | operative time
  measurements of intraoperative heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Lecturer of Anesthesia and Pain Management, National Cancer Institute, Cairo University
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be available upon reasonable request through contacting the principle investigator